CLINICAL TRIAL: NCT05535127
Title: Sequential Strategy of Palpation Plus Ultrasound vs Palpation vs Routine Ultrasound , in Adults for Detection of Cricothyroid Membrane: Protocol of an Adaptive Controlled Randomized Clinical Trial
Brief Title: Sequential Strategy vs Palpation vs Routine Ultrasound for Detection of Cricothyroid Membrane
Acronym: EcoID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IN78-2021
Record Dates: First submitted 2022-05-11; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-03

CONDITIONS: Airway Disease; Intubation; Difficult or Failed; Ultrasound Therapy
MeSH Terms: interventions — Palpation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palpation with " laryngeal handshake" technique " (Active Comparator): With the non-dominant hand, the larynx is stabilized, the hyoid bone is identified with the thumb and index finger by palpation of the greater horns with a horizontal movement from side to side, move thumb and fingers inferiorly to locate thyroid cartilage,Once identified, its location is maintained with the middle finger and thumb, and the index finger travels towards the midline.
  The index finger, already in the midline, makes a longitudinal movement downwards to determine the small depression between the cricoid and thyroid cartilage that corresponds to the cricothyroid membrane.
  Interventions: Diagnostic Test: Palpation with " laryngeal handshake" technique
- Palpation strategy plus sequential ultrasound (Experimental): Palpation is performed with the previously described laryngeal handshake technique If the participant is unable to identify the location of the cricothyroid membrane with certainty, the mixed ultrasound protocol is continued. as decribed in Identification of the cricothyroid membrane with ultrasound
  Interventions: Diagnostic Test: Palpation strategy plus sequential ultrasound
- Identification of the cricothyroid membrane with routine ultrasound (Active Comparator): With the patient on a supine stretcher position, neck extended, with a linear transducer and ultrasound gel, a cross-sectional evaluation of the airway is performed, identifying the cartilaginous referents of the airway. In this case, the midline referent will be the union of the laminae of the thyroid cartilage. The midpoint of the hyperechoic image is located between both referents (MCT).
  Next, tracheal rings are identified, the transducer is moved laterally and a 90° turn is performed for axial evaluation of the MCT. The aim is to preserve the same anatomical landmarks already identified in the transverse plane, the cephalocaudal distance between the thyroid cartilage and the cricoid is evaluated, locating the midpoint with the help of the acoustic shadow generated by a yelco without a needle. Based on these 2 measurements, the topographical location of the MCT will be marked with a visible ink marker under UV light, which will serve as a benchmark for comparison.
  Interventions: Diagnostic Test: Identification of the cricothyroid membrane with routine ultrasound

INTERVENTIONS:
Diagnostic Test: Palpation with " laryngeal handshake" technique — Information alredy included
  Arms: Palpation with " laryngeal handshake" technique "
Diagnostic Test: Palpation strategy plus sequential ultrasound — Information alredy included
  Arms: Palpation strategy plus sequential ultrasound
Diagnostic Test: Identification of the cricothyroid membrane with routine ultrasound — Information alredy included
  Arms: Identification of the cricothyroid membrane with routine ultrasound

SUMMARY:
EcoID is a study designed as an adaptive controlled clinical trial with a first phase of superiority and a second phase of non-inferiority with change of control, of parallel groups, random assignment and blinding of investigators measuring outcome.

DETAILED DESCRIPTION:
Methodology: Methods, techniques and tools provided. Describe the design, study population, materials, procedures and analysis plan:

EcoID is a study designed as an adaptive controlled clinical trial with a first phase of superiority and a second phase of non-inferiority with change of control, of parallel groups, random assignment and blinding of investigators measuring outcome.

A Bayesian statistical approach will be used for the analysis and inferences of the information obtained from the clinical trial. The use of an adaptive study is justified given that there is uncertainty if the sequential strategy is superior to palpation, so performing the sequential experiment optimizes sample collection. In case the intervention does not pass phase 1, it is not necessary to expose more patients to compare the intervention by the second control.

By using a Bayesian statistical approach, it is possible to use the phase 1 sample as a prior probability distribution.

Therefore, the adaptive sample of phase 2 is optimized, achieving the best statistical performance with the least amount of time and resources, benefits found in this type of design The study population will be adult patients of the IPS Universitaria, who accept participation in the study and sign the informed consent.

In phase 1 of the study, a comparison will be made between identification of the MCT by palpation and the intervention of identification by the sequential strategy of palpation plus ultrasound, this consists of an assessment by palpation and in the event that the participant is not sure in the identification advances in ultrasound assessment. A sample of 129 patients is calculated for each arm. The superiority of the intervention over palpatory control will be assessed, only if this superiority is demonstrated will advance to phase 2.

For phase 2, a comparison will be made between identification of the MCT by routine ultrasound and the intervention of identification by the strategy sequential palpation plus ultrasound. The sample will be calculated based on the results of the first phase, the hypothesis will be to demonstrate that this intervention strategy is not inferior to routine ultrasound.

The accuracy of the controls and the intervention will be compared against the ultrasound identification of an airway expert with a CUSUM curve greater than 90%.

Materials:

* Training activities both in MCT identification strategy by palpation with the laryngeal handshake technique, routine ultrasound to achieve a CUSUM curve > 80% in the participants and training in the sequential strategy.
* Mindray M9 ultrasound scanner with linear probe without needle
* Yelco gel -Chronometer
* UV visible ink marker -Black ink marker

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old.
* Acceptance of participation in the clinical study
* Informed consent signature
* Hopitalizated

Exclusion Criteria:

* Patients with tracheostomy or other ventilation devices in the cervical region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of adequate cricothyroid membrane identification by group | through study completion, an average of 30 minutes
  Adequate Identification of the cricothyroid membrane For the present study, it is defined as the concordance between the marking performed by any of the interventions and the marking performed by an expert. This must have a distance of less than 5 mm both in the axial and longitudinal planes. An expert in the field is defined as a professional who works using advanced airway management strategies, and has published on airway ultrasonography and/or performs a CUSUM curve for MCT identification >90%.

SECONDARY OUTCOMES:
Degree of difficulty | 30 minutes
  perceived by evaluators in the identification of the cricothyroid membrane: It is understood as the perception of difficulty of each intervention by the administrators of the intervention.
Time to detection | through study completion, an average of 10 minutes
  Defined as the time from the first contact with the patient by the administrator of the intervention, until the marking of the cricothyroid membrane with any of the interventions
Longitudinal deviation | through study completion, an average of 10 minutes
  Defined as the distance in millimeters between the marking made by the administrator of the intervention and the expert evaluator of the outcome in the lateral plane.
Lateral deviation in mm | through study completion, an average of 10 minutes
  Defined as the distance in millimeters between the marking made by the administrator of the intervention and the expert evaluator of the outcome in the lateral plane.
Participant satisfaction | through study completion, an average of 10 minutes
  Defined as the patients' global perception of satisfaction with the technique.
  For this measurement, a global Likert-type scale will be used, whose score ranges between 1 and 7, with 1 being very dissatisfied and 7 being very satisfied.
Satisfaction of the administrators of the intervention | through study completion, an average of 10 minutes
  Defined as the global perception of satisfaction with the technique by the participants administering the intervention.
  For this measurement, a global Likert-type scale will be used, whose score ranges between 1 and 7, with 1 being very dissatisfied and 7 being very satisfied.
Perception of adherence to the technique | through study completion, an average of 10 minutes
  Defined as the global perception of future use of the technique by the administrators of the intervention.
  For this measurement, a Likert-type global scale will be used, whose score ranges between 1 and 7, with 1 being a very poor perception of use in the future and 7 being a very high perception of use in the future

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Zamudio, Prof, Principal Investigator — mario.zamudio@udea.edu.co
Locations (1):
- Antioquia´s University, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No
public deposit

REFERENCES:
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Jones PM, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Kovacs G; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 1. Difficult airway management encountered in an unconscious patient. Can J Anaesth. 2021 Sep;68(9):1373-1404. doi: 10.1007/s12630-021-02007-0. Epub 2021 Jun 18. PMID 34143394
- [Background] Rai Y, You-Ten E, Zasso F, De Castro C, Ye XY, Siddiqui N. The role of ultrasound in front-of-neck access for cricothyroid membrane identification: A systematic review. J Crit Care. 2020 Dec;60:161-168. doi: 10.1016/j.jcrc.2020.07.030. Epub 2020 Aug 13. PMID 32836091
- [Background] Zanetti G, Mandressi A, Ruoppolo M, Montanari E, Pisani E. Infected renal stones and defects of ureteral peristalsis. Arch Ital Urol Nefrol Androl. 1987 Dec;59(2):71-4. No abstract available. PMID 2976186
- [Background] Altun D, Ali A, Koltka K, Buget M, Celik M, Doruk C, Camci AE. Role of ultrasonography in determining the cricothyroid membrane localization in the predicted difficult airway. Ulus Travma Acil Cerrahi Derg. 2019 Jul;25(4):355-360. doi: 10.14744/tjtes.2019.65250. PMID 31297781